CLINICAL TRIAL: NCT01247129
Title: Delaying the Superficial Inferior Epigastric Artery (SIEA) Flap: A Solution to the Problem of the Small Caliber of the Donor Artery
Brief Title: Delaying the Superficial Inferior Epigastric Artery (SIEA) Flap and Determining the Change in SIEA Diameter and Blood Flow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University Medical Centre Maribor (Other)
Responsible Party: Minja Gregorič, University Medical Centre Maribor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-2010
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Breast Neoplasms
Keywords: Superficial inferior epigastric artery flap, delay phenomenon
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIEA,delay procedure,widening of diameter (Experimental)
  Interventions: Procedure: Delay procedure of SIEA flap.

INTERVENTIONS:
Procedure: Delay procedure of SIEA flap. — Ligating the deep inferior epigastric artery ipsilaterally to the planned raising of the SIEA flap 2 weeks prior to the reconstructive procedure.

SUMMARY:
The purpose of this study is to determine whether delaying the superficial inferior epigastric artery (SIEA) flap results in widening of diameter and enhancing of blood flow of its donor artery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery for lower extremities varicose veins

Exclusion Criteria:

* patients who previously underwent operations of the lower abdomen (abdominoplasty and inguinal hernia repair)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

REFERENCES:
- [Derived] Gregoric M, Flis V, Milotic F, Mrda B, Stirn B, Arnez ZM. Delaying the superficial inferior epigastric artery flap: a solution to the problem of the small calibre of the donor artery. J Plast Reconstr Aesthet Surg. 2011 Sep;64(9):1181-6. doi: 10.1016/j.bjps.2011.04.009. Epub 2011 May 10. PMID 21561823